CLINICAL TRIAL: NCT07241702
Title: The Effect of Hybrid Closed-loop Systems on Markers of Endothelial, Myocardial and Vascular Function in Patients With Type 1 Diabetes.
Brief Title: EFFECT OF HYBRID CLOSED-LOOP SYSTEMS ON CARDIOVASCULAR MARKERS IN TYPE 1 DIABETES.
Status: Active, not recruiting | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, VAIA LAMBADIARI, Professor of Internal Medicine-Endocrinology, Attikon Hospital
Other Study IDs: TYPE 1-HCLS
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HCL group: Patients will recieve hybrid closed loop system
  Interventions: Device: HCLS
- SGLT-2i group: Patients will recieve SGLT-2i as add on treatment to multiple daily injections
  Interventions: Drug: SGLT2 inhibitor
- MDI group: Patients will recieve intensification of MDI treatment.
  Interventions: Drug: MDI

INTERVENTIONS:
Device: HCLS — Hybrid Closed-Loop System treatment
  Groups: HCL group
Drug: SGLT2 inhibitor — SGLT-2 Inhibitor Treatment
  Groups: SGLT-2i group
Drug: MDI — Multiple Daily Injection Insulin treatment
  Groups: MDI group

SUMMARY:
This is a prospective, non-randomized, observational cohort study conducted in adult patients with type 1 diabetes.Participants with poorly controlled T1D under multiple daily injection (MDI) treatment will be assigned to one of three treatment groups:

1. hybrid closed-loop systems (HCLS) or
2. Sodium glucose co-transporter 2 inhibitors (SGLT-2i) added to MDI or
3. intensification of MDI treatment. Markers of endothelial and cardiovascular function will be assessed at baseline, at 6 and 12 months post-treatment. The primary objactive of the study is to evaluate the effect of HCLS on cardiovacular and endothelial function compared to MDI or SGLT-2i in T1D.

DETAILED DESCRIPTION:
Patients with type 1 diabetes mellitus (T1DM) present subclinical signs of vascular and endothelial dysfunction earlier compared to healthy individuals. Hybrid closed loop systems (HCLS) are currently the gold standard method for glycemic management, however, the data regarding its superiority in terms of the prevention of subclinical vascular and endothelial dysfunction are scarce. The aim of this study is to determine whether treatment with HCLS improves vascular and endothelial function compared to multiple daily injections (MDI) or Sodium glucose co-transporter 2 inhibitors (SGLT-2i) in patients with T1DM. Partcipants with poorly controlled T1DM under MDI treatment, will be assigned to receive either:

1. HCLS or
2. SGLT-2i as an add-on treatment to MDI or
3. intensification of MDI treatment.

We will assess at baseline and 6 and 12 months post-treatment:

(i) glycemic parameters derived via continuous glucose monitoring (GGM) (ii) pulse wave velocity (PWV) (iii)central systolic and diastolic blood pressure (cSBP, cDBP) (iv) the perfused boundary region (PBR) of the sublingual arterial microvessels, as a marker of endothelial glycocalyx integrity.

(v) global longitudinal strain(GLS).

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* history of type 1 diabetes with diabetes duration > 5 years
* HbA1c ≥ 7% and ≤ 10%
* eGFR> 60ml/min/1,73m2.

Exclusion Criteria:

* history of malignancy within the last 5 years
* severe hepatic impairment
* cardiovascular events within the recent three months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with poorly controlled type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pulse Wave Velocity | Baseline, Six Months, Twelve months
  The investigators will assess pulse wave velocity as a marker of arterial stiffness at baseline, at six and twelve months post-treatment
Perfused Boundary Region | Baseline, Six Months, Twelve months
  The investigators will assess perfused boundary region as a marker of endothelial glycocalyx integrity at baseline, at six and twelve months post-treatment
Global Longitudinal Strain | Baseline, Six Months, Twelve months
  The investigators will assess global londitudinal strain as a marker of myocardial function at baseline, at six and twelve months post-treatment

SECONDARY OUTCOMES:
Central Systolic Blood Pressure | Baseline, Six Months, Twelve months
  The investigators will assess central systolic blood pressure as a marker of vascular function at baseline, at six and twelve months post-treatment
Central Diastolic Blood Pressure | Baseline, Six Months, Twelve months
  The investigators will assess central diastolic blood pressure as a marker of vascular function at baseline, at six and twelve months post-treatment
Augmentation Index | Baseline, Six Months, Twelve months
  The investigators will assess Augmentation Index as a marker of vascular function at baseline, at six and twelve months post-treatment
Flow mediated dilation | Baseline, Six Months, Twelve months
  The investigators will assess Flow Mediated Dilation as a marker of endothelial function at baseline, at six and twelve months post-treatment
Coronary flow reserve | Baseline, Six Months, Twelve months
  The investigators will assess Coronary flow reserve at baseline, at six and twelve months post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon University General Hospital, Athens, Greece